CLINICAL TRIAL: NCT05790265
Title: Assessing Innovative Wireless and Wearable Sensors for Continuous Blood Pressure Measurement in Obese and Super-obese Pregnant Women
Brief Title: Assessing Innovative Wireless and Wearable Sensors for Continuous Blood Pressure Measurement in Obese Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sibel Health Inc. (Industry)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-2375
Record Dates: First submitted 2023-03-15; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Comparison of ANNE One system blood pressure measurements to arterial line (Experimental)
  Interventions: Device: ANNE One

INTERVENTIONS:
Device: ANNE One — Chest sensor for single lead ECG and finger sensor for pulse oximetry.

SUMMARY:
This study is a prospective study targeting at least 20 obese and super-obese patients admitted to Labor & Delivery (L&D) for delivery at UNC Medical Center. Patients with clinical indicated radial A-lines either planned or already in-situ will be offered participation. The study will evaluate the accuracy of noninvasive blood pressure measurements with the ANNE One system to blood pressure readings with the radial A-line.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Ability and willingness to provide written informed consent
* Admitted for delivery at UNC Medical Center
* BMI of >= 40 kg/m2
* Clinically indicated radial A-lines either planned or already in-situ prior to delivery

Exclusion Criteria:

* Skin sensitivity or allergy that precludes placement of ANNE One
* Any condition (social or medical) which, in the opinion of the study staff would make any study participation unsafe or complicate data interpretation
* Expected delivery within <= 1 hour of arrival to L&D

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean absolute error (MAE) and standard deviation of blood pressure measurements with ANNE One compared to arterial line | 8 hours
  Mean absolute error and standard deviation between the non-invasive blood pressure measurement provided by the device under test and the invasive blood pressure measurement from the arterial line.